CLINICAL TRIAL: NCT04135599
Title: Transcranial Direct Current Stimulation of the Bilateral Dorsolateral Prefrontal Cortex for Alcohol Use Disorders: A Randomised, Sham-controlled Clinical Trial
Brief Title: A Study of the Effectiveness of Direct Current Stimulation for Alcohol Use Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NZhong-004
Record Dates: First submitted 2019-09-28; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Active Comparator): Participants received 1.5mA tDCS for 20 minutes in 10 consecutive days.
  Interventions: Device: transcranial direct current stimulation
- sham tDCS (Sham Comparator): Participants received sham tDCS for 20 minutes in 10 consecutive days.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a non-invasive, safe and easy-to-operate neuro-electrophysiological technique, which becoming an emerging therapeutic option for many mental disorders.It can modulate cortical excitability of target brain region, neuron plasticity and brain connections. Previous studies suggest that tDCS could reduce cue-induced craving and improve cognition in drug addiction.

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive, safe and easy-to-operate neuro-electrophysiological technique, which becoming an emerging therapeutic option for many mental disorders.It can modulate cortical excitability of target brain region, neuron plasticity and brain connections. Previous studies suggest that tDCS could reduce cue-induced craving in drug addiction.

Objective:In this study, the investigators employed real and sham tDCS of the bilateral dorsolateral prefrontal cortex (DLPFC) to test the effect of whether it could reduce cue-induced craving, influence cognitive function in alcoholics and explore its underlying mechanism with functional magnetic resonance imaging (fMRI).

Methods: The investigators perform a randomized sham-controlled study in which 40 inpatient alcoholics will be randomized to receive 10 sessions of 20min sham or 1.5mA tDCS to the bilateral DLPFC (anodal right/cathodal left). The neuroimaging data, craving after exposed to alcohol-associated cues and the cognition task at baseline and after stimulation will be collected.

The investigators hypothesized that tDCS stimulating the DLPFC decreases cue-induced craving and improves cognition, which might be associated with the functional connectivity alterations.

ELIGIBILITY:
Inclusion Criteria:(1)Clinical diagnosis of severe AUD defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth edition (DSM-5); (2)Must be able to look and hear; (3) Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) score less than 10.

Exclusion Criteria:(1) Clinical diagnosis of substance use disorder other than an alcohol or nicotine use disorder defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth edition (DSM-5)；(2) Severe brain injury, stroke, seizure, epilepsy or other major neurological diseases ; (3) Schizophrenia, bipolar disorder, depression or other Axis I disorder of DSM-V criteria;(4)any contraindication for fMRI scanning.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline functional magnetic resonance imaging at 2 weeks | Two weeks
  Stop signal task during fMRI scanning (Philips Ingenia 3.0T MRI).

SECONDARY OUTCOMES:
cue-induced craving | Two weeks
  Participants were instructed to pay close attention to real alcoholic beverages and rate their level of craving after smelling and recalling the last time they engaged in alcohol use. Craving was assessed by visual analog scales (VAS), with 0 mm being "no craving"and 100 mm representing "most craving ever experienced for alcohol".
Cognitive function | Two weeks
  Chinese version of the CogState Battery was used to assess cognitive function. We selected two tasks: Two back task (working memory) and Identification task (attention) which were displayed on a green screen with standardized instructions before each task beginning.The accuracy in Two back task and the speed in Identification task are our focus.
Relapse | One month after discharge from the hospital
  Meet the criteria for mild to severe AUD defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth edition (DSM-5)

CONTACTS AND LOCATIONS:
Overall Officials: Na Zhong, Doctor, Principal Investigator — Shanghai Mental Health Center